CLINICAL TRIAL: NCT02653794
Title: The Variations of Macular Thickness in Juvenile Subjects With Mild-to-Moderate Refractive Error
Brief Title: The Variations of Macular Thickness in Juvenile Subjects
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Erping Long, Medical doctor,Childhood Cataract Program of the Chinese Ministry of Health(CCPMOH), Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: CCPMOH2016-China1
Record Dates: First submitted 2016-01-10; First posted 2016-01-12 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Cataract;Macular Thickness
Keywords: Juvenile Subjects'characteristics

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
It is reported that it takes a period form 22 weeks pregnant to the first 45 months of life for macular region to develop from structural formation to functional integrity. However, children are still in the critical period of plastic visual development, for their visual acuity has not yet reached the level of adults. Similarly macular retinal structure may develop with age. It is very important to study in macular thickness of this period and to have a proper cognition of it and the relation between macular thickness and other ocular parameter for the research of retinal development and diseases and the early screen of fundus diseases.

DETAILED DESCRIPTION:
It is reported that it takes a period form 22 weeks pregnant to the first 45 months of life for macular region to develop from structural formation to functional integrity. However, children are still in the critical period of plastic visual development, for their visual acuity has not yet reached the level of adults. Similarly macular retinal structure may develop with age. It is very important to study in macular thickness of this period and to have a proper cognition of it and the relation between macular thickness and other ocular parameter for the research of retinal development and diseases and the early screen of fundus diseases.

Optical Coherence Tomography (OCT) is an imaging technique widely used in clinic in last twenty years. According to the base theory of dim coherent light interference machine, OCT detect the back-reflection or scattering signal of biological tissue to the incident dim coherent light, and acquire the two-dimension or three- dimension image of biological tissue by scan. It enables the characteristic of tissue's microstructure in vivo and makes it possible to observe dynamically developing process of diseases so that it has become an essential test for macular and optic nerve diseases with unmatched measurement reproducibility. It also enables high-resolution and noninvasive imaging of the retinal lamina, the organizational structure of macular. It is most often used clinically to demonstrate the macular morphology, treatment response and disease progression clinically. However, who researchers studyed in through OCT were mostly patients with retinal disease and adults. There was few study focused on OCT's application to children.

In this study, the investigators aims to measure macular thickness (MT) using spectral-domain optical coherence tomography (SD-OCT) and to investigate MT variations with sex, age, laterality, refraction error (RE) and axial length (AL).

ELIGIBILITY:
Inclusion Criteria:

* age from 4 to 17 years
* children with the mild-to-moderate refraction error(from 0 to -6.00D)

Exclusion Criteria:

* children with visual complaints

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects consisted of Zhongshan Ophthalmic Center (ZOC) and Hualong Primary School (HPS)), who came from ZOC group were mild-to-moderate refraction error while who come from HPS group had no visual complaints.
Sampling Method: Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
change of Macular thickness | 4 to 17 years after birth
  MT measurement using SD-OCT(an imaging technique widely used in clinic in last twenty years)
change of axis length measurement using an IOLMaster | 4 to 17 years after birth
  axis length measurement using an IOLMaster

CONTACTS AND LOCATIONS:
Overall Officials: Erping Long, M.D.,Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Yizhi Liu, M.D.;Ph.D., Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University; Haotian Lin, M.D.;Ph.D., Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Ojaimi E, Rose KA, Smith W, Morgan IG, Martin FJ, Mitchell P. Methods for a population-based study of myopia and other eye conditions in school children: the Sydney Myopia Study. Ophthalmic Epidemiol. 2005 Feb;12(1):59-69. doi: 10.1080/09286580490921296. PMID 15848921
- [Background] Wakitani Y, Sasoh M, Sugimoto M, Ito Y, Ido M, Uji Y. Macular thickness measurements in healthy subjects with different axial lengths using optical coherence tomography. Retina. 2003 Apr;23(2):177-82. doi: 10.1097/00006982-200304000-00007. PMID 12707596
- [Background] Chen S, Wang B, Dong N, Ren X, Zhang T, Xiao L. Macular measurements using spectral-domain optical coherence tomography in Chinese myopic children. Invest Ophthalmol Vis Sci. 2014 Oct 14;55(11):7410-6. doi: 10.1167/iovs.14-13894. PMID 25316719
- [Background] Lim MC, Hoh ST, Foster PJ, Lim TH, Chew SJ, Seah SK, Aung T. Use of optical coherence tomography to assess variations in macular retinal thickness in myopia. Invest Ophthalmol Vis Sci. 2005 Mar;46(3):974-8. doi: 10.1167/iovs.04-0828. PMID 15728555
- See also: Description Home page of Zhongshan Ophthalmic Center — http://www.gzzoc.com/